CLINICAL TRIAL: NCT04247542
Title: ACX-362E [Ibezapolstat] for Oral Treatment of Clostridioides Difficile Infection: A Phase 2A Open-Label Segment Followed by a Phase 2B Double-Blind Vancomycin-Controlled Segment
Brief Title: ACX-362E [Ibezapolstat] for Oral Treatment of Clostridioides Difficile Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acurx Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACX-362E-201
Record Dates: First submitted 2020-01-23; First posted 2020-01-30 (Actual); Results first posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Clostridium Difficile Infection
Keywords: Clostridioides difficile; CDAD (Clostridioides difficile-associated diarrhea); DNA polymerase IIIC
MeSH Terms: conditions — Clostridium Infections | interventions — Ibezapolstat; Vancomycin

STUDY DESIGN:
Intervention Model Description: In Segment 2B, approximately 64 patients will be randomly assigned in a 1:1 fashion to ibezapolstat or the standard of care positive control, vancomycin.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Vancomycin capsules will be over-encapsulated to have identical appearance to ibezapolstat capsules. Placebo capsules will be used to enable a double-dummy, double-blind design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ibezapolstat (Experimental): Active investigational antibacterial agent: ibezapolstat 450 mg po Q12H x 10 days
  Interventions: Drug: Ibezapolstat
- Vancomycin (Active Comparator): Standard of care: Vancomycin 125 mg po Q6H x 10 days
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Ibezapolstat — Investigational antibacterial agent
  Other Names: ACX-362E
  Arms: Ibezapolstat
Drug: Vancomycin — Active comparator
  Other Names: Vancomycin oral
  Arms: Vancomycin

SUMMARY:
Segments 2A and 2B of this trial evaluate the safety, efficacy, pharmacokinetics, fecal concentrations, and fecal microbiome effects of ACX-362E [ibezapolstat] in patients with C. difficile infection (CDI).

DETAILED DESCRIPTION:
This Phase 2, multicenter, open-label single-arm segment (2A) followed by a double-blind, randomized, active-controlled segment (2B) is designed to evaluate ACX-362E in the treatment of CDI. Segment 2A of this trial was an open-label study of up to 20 patients at 6 study centers and was terminated early at 10 patients based on the protocol-specified Trial Oversight Committee's assessment of the compelling efficacy and safety data. Patients were treated with 450 mg of oral ibezapolstat twice daily for 10 days. The trial will advance to Segment 2B which is a double-blind comparison of ibezapolstat to the standard of care, oral vancomycin, in approximately 64 subjects (1-1 randomization) at up to approximately 15 sites.

Subjects will be evaluated for cure, safety, and tolerability. All subjects in both segments will have stool samples tested for microbiome profiles. Pharmacokinetic (PK) testing for systemic exposure will be performed on blood samples. Stool samples will be tested for study drug concentration.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 to 90 years of age, inclusive, at the time of Screening.
2. Capable of reading, understanding, and signing the written informed consent; able to adhere to all study procedures and attend all scheduled study visits.
3. Confirmed diagnosis of mild or moderate CDI as defined by the Infectious Diseases Society of America/Society for Healthcare Epidemiology of America guidelines (McDonald et al. 2018). Subjects will be diagnosed with CDI based on clinical and laboratory findings:

   1. The presence of diarrhea, defined as passage of ≥ 3 UBMs within 24 hours before dosing; an unformed stool is defined as a Type 5, 6, or 7 on the Bristol Stool Chart (Appendix 2)
   2. A stool test result positive for the presence of C. difficile free toxins using tests that detect toxin A/B (and it is prospectively agreed with the Sponsor). The Sponsor will provide a toxin A/B test kit if the site does not have it as part of standard of care test.
   3. Mild or moderate CDI as defined as a white blood cell count of ≤ 15000 cells/mL and a serum creatinine level < 1.5 mg/dL.

Exclusion Criteria:

1. Received more than 24 hours of dosing (> 4 doses) of oral vancomycin for the current episode of CDI before first dose of study drug.
2. Received more than 24 hours of dosing (> 2 doses) of oral fidaxomicin for the current episode of CDI before first dose of study drug.
3. Received more than 24 hours of dosing (> 3 doses) of oral/IV metronidazole for the current episode of CDI before first dose of study drug.
4. Received any other antibacterial therapy for the current CDI episode within 48 hours before the first dose of study drug.
5. Subjects considered treatment failures on prior antibiotics for their current episode of CDI will be excluded.
6. More than 3 episodes of CDI in the previous 12 months or more than 1 prior episode in the last 3 months, excluding the current episode.
7. Severe, complicated, or life-threatening fulminant CDI with evidence of hypotension (systolic blood pressure less than 90 mmHg), septic shock, peritoneal signs or ileus, or toxic megacolon.
8. Elevated liver transaminases (alanine aminotransferase [ALT], aspartate aminotransferase [AST]) greater than 2 times ULN.
9. Active inflammatory bowel disease (Crohn's disease, ulcerative colitis, Irritable Bowel Syndrome with chronic diarrhea).
10. Any other non-C. difficile diarrhea.
11. Active gastroenteritis because of Salmonella, Shigella, Escherichia coli 0157H7, Yersinia or Campylobacter, a parasite, or virus within the past 2 weeks.
12. Had a known positive diagnostic test for other relevant gastrointestinal [GI] pathogens in the 2 weeks before study drug treatment and/or colonization/infection by ova or parasites.
13. Major GI surgery (ie, significant bowel resection) within 3 months of enrollment (does not include appendectomy or cholecystectomy).
14. Prior or current use of anti-C. difficile toxin antibodies.
15. Have received a vaccine against C. difficile or its toxins.
16. Anticipated that systemic antibacterial therapy for a non-CDI infection will be required for > 7 days after start of study therapy.
17. Actively taking anti-diarrheals, and unable to discontinue anti-diarrheal medication, or any medication with the potential to slow bowel movement (for opiates, a stable dose, including use as needed, is permitted).
18. Actively taking Saccharomyces boulardii and unwilling to discontinue during the study period.
19. Received a fecal transplant in the previous 3 months.
20. Received laxatives in the last 48 hours.
21. Unable or unwilling to stop taking oral probiotics for the duration of the study.
22. Received intravenous immunoglobulin within 3 months before study drug treatment.
23. Sepsis.
24. Have a known current history of significantly compromised immune system such as:

    1. Subjects with a known history of human immunodeficiency virus infection and CD4 <200 cells/mm3 within 6 months of start of study therapy.
    2. Severe neutropenia with neutrophil count < 500 cells/mL.
    3. Concurrent intensive induction chemotherapy, radiotherapy, or biologic treatment for active malignancy.
25. Pregnant or lactating women.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Silverman, MD, Study Director — Acurx Pharmaceuticals Inc.
Locations (29):
- United States (29):
  - Acurx Site #118: Dr Janet Reiser, Scottsdale, Arizona
  - Acurx Site #115: Dr Neera Grover, Apple Valley, California
  - Acurx Site #125: Dr Karen Simon, Camarillo, California
  - Acurx Site #111: Dr Jatinder Pruthi, Lancaster, California
  - Acurx Site #131: Dr Michael Jardula, Palm Springs, California
  - Acurx Site #129: Dr Stuart Cohen, Sacramento, California
  - Acurx Site #105, Doral, Florida
  - Acurx Site #122: Dr Faride Ramos, Doral, Florida
  - Acurx Site #101: Dr Idalia Acosta, Miami, Florida
  - Acurx Site #124: Dr Yunior Silva-Barrero, Miami, Florida
  - Acurx Site #108: Dr Idania Garcia Del Sol, Miami, Florida
  - Acurx Site #116: Dr Erick Juarez, Miami, Florida
  - Acurx Site #119: Dr Jorge Paoli-Bruno, Miami, Florida
  - Acurx Site #107: Dr Belkis Delgado, Miami Springs, Florida
  - Acurx Site #117: Dr Rafael Companioni, Panama City, Florida
  - Acurx Site #102: Dr Richard Nathan, Idaho Falls, Idaho
  - Acurx Site #123: Dr Harry Schrager, Newton, Massachusetts
  - Acurx Site #104: Dr JeanMarie Houghton, Worcester, Massachusetts
  - Acurx Site #103: Dr John Pullman, Butte, Montana
  - Acurx Site #130: Dr Michael DiGiovanna, North Massapequa, New York
  - Acurx Site #127: Dr Christopher Connolley, Winston-Salem, North Carolina
  - Acurx Site #126: Dr Andrew Pearson, Myrtle Beach, South Carolina
  - Acurx Site #114: Dr Eugene Ryan, Chattanooga, Tennessee
  - Acurx Site #121: Dr Ramesh Gowrappala, Houston, Texas
  - Acurx Site #120: Dr Vanna Gold, Lampasas, Texas
  - Acurx Site #113: Dr Jennifer Vincent, Temple, Texas
  - Acurx Site #110: Dr Val Hansen, Bountiful, Utah
  - Acurx Site #106: Dr Bezawit Tekola, Fairfax, Virginia
  - Acurx Site #109: Dr Robert Brennan, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xu WC, Silverman MH, Yu XY, Wright G, Brown N. Discovery and development of DNA polymerase IIIC inhibitors to treat Gram-positive infections. Bioorg Med Chem. 2019 Aug 1;27(15):3209-3217. doi: 10.1016/j.bmc.2019.06.017. Epub 2019 Jun 11. PMID 31221610
- [Background] Dvoskin S, Xu WC, Brown NC, Yanachkov IB, Yanachkova M, Wright GE. A novel agent effective against Clostridium difficile infection. Antimicrob Agents Chemother. 2012 Mar;56(3):1624-6. doi: 10.1128/AAC.06097-11. Epub 2011 Dec 27. PMID 22203600
- [Background] Garey KW, Begum K, Lancaster C, Gonzales-Luna A, Bui D, Mercier J, Seng Yue C, Ducharme MP, Hu M, Vince B, Silverman MH, Alam MJ, Kankam M. A randomized, double-blind, placebo-controlled, single and multiple ascending dose Phase 1 study to determine the safety, pharmacokinetics and food and faecal microbiome effects of ibezapolstat administered orally to healthy subjects. J Antimicrob Chemother. 2020 Dec 1;75(12):3635-3643. doi: 10.1093/jac/dkaa364. PMID 32892222
- [Result] Garey KW, McPherson J, Dinh AQ, Hu C, Jo J, Wang W, Lancaster CK, Gonzales-Luna AJ, Loveall C, Begum K, Jahangir Alam M, Silverman MH, Hanson BM. Efficacy, Safety, Pharmacokinetics, and Microbiome Changes of Ibezapolstat in Adults with Clostridioides difficile Infection: A Phase 2a Multicenter Clinical Trial. Clin Infect Dis. 2022 Sep 30;75(7):1164-1170. doi: 10.1093/cid/ciac096. PMID 35134880
- [Result] Eubank TA, Alam MJ, Begum K, McPherson JK, Jo J, Silverman MH, and Garey KW. A phase 2b, randomized double-blind study of ibezapolstat compared with vancomycin for the treatment of C. difficile infection: clinical and microbiome evaluation. Poster session presented at: IDWeek 2024; 2024 October 16-19; Los Angeles, CA.
- [Result] Garey KW, Alam MJ, Begum K, McPherson JK, Eubank TA, Jo J, and Silverman MH. Microbiome Results from the phase 2, randomized, double-blind study of ibezapolstat compared with vancomycin for the treatment of Clostridioides difficile infection. Slide presentation at: 8th International Clostridioides difficile Symposium; 2024 September 17-19; Bled, Slovenia.
- [Derived] Eubank TA, Jo J, Alam MJ, Begum K, McPherson JK, Le TM, Horvath TD, Haidacher SJ, Poggio EC, Lin R, Yue CS, Ducharme MP, Koudssi G, Mercier J, Alder JD, Silverman MH, Garey KW; Ibezapolstat Phase 2 Investigator Group. Efficacy, safety, pharmacokinetics, and associated microbiome changes of ibezapolstat compared with vancomycin in adults with Clostridioides difficile infection: a phase 2b, randomised, double-blind, active-controlled, multicentre study. Lancet Microbe. 2025 Aug;6(8):101126. doi: 10.1016/j.lanmic.2025.101126. Epub 2025 Jun 11. PMID 40516571
- See also: Sponsor website-Acurx Pharmaceuticals — http://www.acurxpharma.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Segment 2A, Ibezapolstat Open-Label Arm: 14 enrolled. Segment 2B, Vancomycin-Controlled Double-Blind: 39 enrolled.
Pre-assignment Details: Segment 2A: 4 participants failed screening. 10 participants proceeded to treatment. Segment 2A participants did not participate in Segment 2B.
  Segment 2B: 7 participants failed screening. 32 participants proceeded to randomization and treatment. Segment 2B did not include Segment 2A participants.
Groups:
- Segment 2A: Ibezapolstat (ACX-362E) Open-Label Single-Arm: Participants with diarrhea caused by C. difficile were treated with ibezapolstat 450 mg orally (3 x 150 mg capsules) every 12 hours for 10 days. Study drug was administered with 240 mL water. Participants were followed for recurrence for 28±2 days, regardless of response to ibezapolstat. Safety, tolerability, and efficacy were assessed by the Trial Oversight Committee which then recommended early termination of this segment of the trial and advancement to the 2B Segment because the first 10 patients demonstrated clinical cure.
- Segment 2B: Ibezapolstat Arm--Double-blind, Randomized, Active-controlled Clinical Segment: Participants with diarrhea caused by C. difficile who were randomized to this arm received 450 mg ibezapolstat (3 x 150 mg capsules) every 12 hours for 10 days with placebo every 12 hours for 10 days (to maintain blind). Participants were followed for 28±2 days for recurrence. Blinding was maintained by over-encapsulation.
- Segment 2B: Vancomycin Arm--Double-blind, Randomized, Active-controlled Clinical Segment: Participants with diarrhea caused by C. difficile who were randomized to this arm received vancomycin every 6 hours (1 capsule 125 mg + 2 placebo capsules every 12 hours or 1 capsule 125 mg every 12 hours). Participants were followed for 28±2 days for recurrence. Blinding was maintained by over-encapsulation.
Period: 2A: Ibezapolstat Open-Label Single-Arm
Arm/Group | Segment 2A: Ibezapolstat (ACX-362E) Open-Label Single-Arm | Segment 2B: Ibezapolstat Arm--Double-blind, Randomized, Active-controlled Clinical Segment | Segment 2B: Vancomycin Arm--Double-blind, Randomized, Active-controlled Clinical Segment
Started (Segment 2B did not start until after Segment 2A was completed.) | 10 | 0 | 0
Completed | 10 | 0 | 0
Not Completed | 0 | 0 | 0
Period: 2B: Double-Blind Active-Controlled
Arm/Group | Segment 2A: Ibezapolstat (ACX-362E) Open-Label Single-Arm | Segment 2B: Ibezapolstat Arm--Double-blind, Randomized, Active-controlled Clinical Segment | Segment 2B: Vancomycin Arm--Double-blind, Randomized, Active-controlled Clinical Segment
Started (Segment 2A participants did not proceed to Segment 2B.) | 0 | 18 | 14
Completed | 0 | 16 | 13
Not Completed | 0 | 2 | 1
Not completed — Did not receive study drug | 0 | 1 | 0
Not completed — Treatment completed but incorrectly recorded as discountinued. | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Segment 2A: Ibezapolstat (ACX-362E) Open-Label Single-Arm | Segment 2B: Ibezapolstat Arm--Double-blind, Randomized, Active-controlled Clinical Segment | Segment 2B: Vancomycin Arm--Double-blind, Randomized, Active-controlled Clinical Segment | Total
Number analyzed (Participants) | 10 | 18 | 14 | 42
Age, Continuous [Mean (Full Range); unit: years] — Population: Segment 2A participants did not participate in Segment 2B. Segment 2B took place after Segment 2A was completed.
  years
    Segment 2A: number analyzed (Participants) | 10 | 0 | 0 | 10
    Segment 2A | 49.5 [27 to 75] |  |  | 49.5 [27 to 75]
    Segment 2B: number analyzed (Participants) | 0 | 18 | 14 | 32
    Segment 2B |  | 63.2 [39 to 83] | 61.8 [49 to 86] | 59.4 [39 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 15 | 11 | 31
  Male | 5 | 3 | 3 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 12 | 11 | 31
  Not Hispanic or Latino | 2 | 6 | 3 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 10 | 18 | 13 | 41
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Segment 2A: Clinical Cure (CC) of Clostridioides Difficile Infection (CDI) Per Protocol (PP)/Modified Intent-to-Treat (mITT) Population
Description: Percentage of patients with CC at the test of cure (TOC) visit on day 12. CC was defined as survival and the resolution of diarrhea in the 24-hour period immediately before end of treatment (EOT--day 10) that was maintained for 48 hours post EOT without a requirement for additional CDI treatment. Diarrhea was defined as 3 or more unformed bowel movements (UBMs) in a 24-hour period; fewer than 3 UBMs was considered as resolution of diarrhea. A UBM was defined as a Type 5, 6, or 7 bowel movement on the Bristol Stool Chart.
Time Frame: 12 days
Population: 10 participants were analyzed in the modified Intent-to-Treat (mITT) and Per Protocol (PP) populations. The mITT population includes all subjects who were treated and assessed at the TOC visit. The PP population consists of patients in the mITT population with no major protocol deviations.
Measure: Count of Participants; unit: Participants
Arm/Group | Segment 2A: Ibezapolstat (ACX-362E) Open-Label Single-Arm
Number analyzed (Participants) | 10
Participants
  CC at TOC, yes | 10
  CC at TOC, no | 0

2. Primary Outcome: Segment 2B Per Protocol (PP) Population: Clinical Cure (CC) of Clostridioides Difficile Infection (CDI)
Description: as for outcome 1
Time Frame: 12 days
Population: PP participants were those in the ITT population who had no major protocol deviations. The ITT population is defined as all randomized subjects, analyzed according to their randomized treatment assignment.
Measure: Count of Participants; unit: Participants
Arm/Group | Segment 2B: Ibezapolstat Arm--double-blind, Randomized, Active-controlled Clinical Segment | Segment 2B: Vancomycin Arm--double-blind, Randomized, Active-controlled Clinical Segment
Number analyzed (Participants) | 16 | 14
Participants
  CC at TOC, yes | 15 | 14
  CC at TOC, no | 1 | 0

3. Primary Outcome: Segment 2B Intent-to-Treat (ITT) Population: Clinical Cure (CC) of Clostridioides Difficile Infection (CDI)
Description: as for outcome 1
Time Frame: 12 days
Population: ITT population is defined as all randomized subjects, analyzed according to their randomized treatment assignment.
Measure: Count of Participants; unit: Participants
Arm/Group | Segment 2B: Ibezapolstat Arm--double-blind, Randomized, Active-controlled Clinical Segment | Segment 2B: Vancomycin Arm--double-blind, Randomized, Active-controlled Clinical Segment
Number analyzed (Participants) | 18 | 14
Participants
  CC at TOC, yes | 15 | 14
  CC at TOC missing | 1 | 0
  CC at TOC, no | 2 | 0

4. Secondary Outcome: Segment 2A: Sustained Clinical Cure (SCC) of Clostridioides Difficile Infection (CDI) Per Protocol (PP)/Modified Intent-to-Treat (mITT) Population
Description: Clinical cure (CC) at the test of cure (TOC) visit (ie, at least 48 hours after end of treatment [day 10]) and no recurrence within 28 days. Recurrence was defined as a new episode of diarrhea (3 or more UBMs in a 24-hour period) with a positive toxin result, using a Sponsor-approved C. difficile free toxin test and, in the opinion of the Investigator, requiring retreatment with an antibacterial agent for C. difficile.
Time Frame: 38 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Segment 2A: Ibezapolstat (ACX-362E) Open-Label Single-Arm
Number analyzed (Participants) | 10
Participants
  SCC, yes | 10
  SCC, no | 0

5. Secondary Outcome: Segment 2B Per Protocol (PP) Population: Sustained Clinical Cure (SCC) of Clostridioides Difficile Infection (CDI)
Description: as for outcome 4
Time Frame: 38 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Segment 2B: Ibezapolstat Arm--double-blind, Randomized, Active-controlled Clinical Segment | Segment 2B: Vancomycin Arm--double-blind, Randomized, Active-controlled Clinical Segment
Number analyzed (Participants) | 16 | 14
Participants
  SCC, yes | 15 | 12
  SCC, no | 1 | 2

6. Secondary Outcome: Segment 2B Intent-to-Treat (ITT) Population: Sustained Clinical Cure (SCC) of Clostridioides Difficile Infection (CDI)
Description: as for outcome 4
Time Frame: 38 days
Population: ITT population is defined as all randomized subjects, analyzed according to their randomized treatment assignment.
Measure: Count of Participants; unit: Participants
Arm/Group | Segment 2B: Ibezapolstat Arm--double-blind, Randomized, Active-controlled Clinical Segment | Segment 2B: Vancomycin Arm--double-blind, Randomized, Active-controlled Clinical Segment
Number analyzed (Participants) | 18 | 14
Participants
  SCC, yes | 15 | 12
  SCC missing | 1 | 0
  SCC, no | 2 | 2

7. Secondary Outcome: Segment 2A: Pharmacokinetics and Systemic Exposure to Ibezapolstat (ACX-362E), Plasma Concentrations
Description: Plasma ibezapolstat concentrations were measured at specified day and time points following dose administration. Amount listed as zero not included in determination of Geometric Mean and CV%.
Time Frame: Days 1, 5, and 10: 2 and 4 hours post-dose
Population: 3 participants from the original population did not have plasma samples taken and were not included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Segment 2A: Ibezapolstat (ACX-362E) Open-Label Single-Arm
Number analyzed (Participants) | 7
ng/mL
  Day 1 Hour 2 | 114.32 (249)
  Day 1 Hour 4 | 305.94 (171)
  Day 5 Hour 2 | 185.37 (244)
  Day 5 Hour 4 | 472.54 (48.0)
  Day 10 Hour 2 | 152.02 (227)
  Day 10 Hour 4 | 527.10 (51.9)

8. Secondary Outcome: Segment 2B: Pharmacokinetics and Systemic Exposure to Ibezapolstat (ACX-362E), Plasma Concentrations
Description: as for outcome 7
Time Frame: Days 1 and 5: 2 and 4 hours post-dose
Population: 3 participants from the original population did not have plasma samples taken and were not included. 1 participant from the original population did not receive the study drug and was not included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Segment 2B: Ibezapolstat Arm--Double-blind, Randomized, Active-controlled Clinical Segment
Number analyzed (Participants) | 14
ng/mL
  Day 1 Hour 2 | 454.82 (178)
  Day 1 Hour 4 | 268.07 (128)
  Day 5 Hour 2 | 441.39 (206)
  Day 5 Hour 4 | 358.52 (151)

9. Secondary Outcome: Segment 2A: Pharmacokinetics and Systemic Exposure to Ibezapolstat (ACX-362E), Fecal Concentrations
Description: Fecal ibezapolstat concentrations were measured for specified days following dose administration. Specified days were 3, 5, 8, 10, 12, 20, and 38. Amount listed as zero not included in determination of Geometric Mean and CV%.
Time Frame: Days -2, 3, 5, 8,10, 12, 20, 30, and 38
Population: Participants with undetectable concentrations were not included in the data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/g
Arm/Group | Segment 2A: Ibezapolstat (ACX-362E) Open-Label Single-Arm
Number analyzed (Participants) | 7
µg/g
  Day -2 | NA (NA) — The measured amount was less than two observed concentration values greater than the lower limit of quantitation (LLOQ). The LLOQ is equal to 2.5 µg/g.
  Day 3 | 285.88 (1058)
  Day 5 | 532.96 (1034)
  Day 8: number analyzed (Participants) | 6
  Day 8 | 943.87 (410)
  Day 10: number analyzed (Participants) | 6
  Day 10 | 1565.77 (271)
  Day 12: number analyzed (Participants) | 6
  Day 12 | 264.47 (1001)
  Day 20: number analyzed (Participants) | 6
  Day 20 | 53.52 (18317)
  Day 30: number analyzed (Participants) | 6
  Day 30 | NA (NA) — The measured amount was less than two observed concentration values greater than the lower limit of quantitation (LLOQ). The LLOQ is equal to 2.5 µg/g.
  Day 38: number analyzed (Participants) | 6
  Day 38 | 267.73 (24)

10. Secondary Outcome: Segment 2B: Pharmacokinetics and Systemic Exposure to Ibezapolstat (ACX-362E), Fecal Concentrations
Description: Fecal ibezapolstat concentrations were measured for specified days following dose administration. Specified days were 3, 5, 8, 10, 12, and 20. Amount listed as zero not included in determination of Geometric Mean and CV%.
Time Frame: Days -2, 3, 5, 8,10,12, 20, 30, and 38
Population: Participants with undetectable concentrations were not included in the data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/g
Arm/Group | Segment 2B: Ibezapolstat Arm--Double-blind, Randomized, Active-controlled Clinical Segment
Number analyzed (Participants) | 12
µg/g
  Day -2: number analyzed (Participants) | 10
  Day -2 | NA (NA) — The measured amount was less than two observed concentration values greater than the lower limit of quantitation (LLOQ). The LLOQ is equal to 2.5 µg/g.
  Day 3 | 411.4 (151)
  Day 5: number analyzed (Participants) | 9
  Day 5 | 407.65 (217)
  Day 8: number analyzed (Participants) | 8
  Day 8 | 716.21 (148)
  Day 10: number analyzed (Participants) | 6
  Day 10 | 958.15 (169)
  Day 12 | 250.52 (63.1)
  Day 20: number analyzed (Participants) | 7
  Day 20 | 12.74 (91.2)
  Day 30: number analyzed (Participants) | 9
  Day 30 | NA (NA) — The measured amount was less than two observed concentration values greater than the lower limit of quantitation (LLOQ). The LLOQ is equal to 2.5 µg/g.
  Day 38: number analyzed (Participants) | 8
  Day 38 | NA (NA) — The measured amount was less than two observed concentration values greater than the lower limit of quantitation (LLOQ). The LLOQ is equal to 2.5 µg/g.

11. Other Pre Specified Outcome: Segment 2A: Time to Resolution of Diarrhea
Description: Time in days from outset of treatment to the first formed bowel movement not followed within the next 24 hours by an unformed bowel movement (UBM), defined as a Type 5, 6, or 7 bowel movement on the Bristol Stool Chart.
Time Frame: 10 days
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days to resolution of diarrhea
Arm/Group | Segment 2A: Ibezapolstat (ACX-362E) Open-Label Single-Arm
Number analyzed (Participants) | 10
Days to resolution of diarrhea | 5 [3 to 7]

12. Other Pre Specified Outcome: Segment 2B: Time to Resolution of Diarrhea
Description: as for outcome 11
Time Frame: 40 days
Population: The Per Protocol (PP) population is represented here. PP participants were those in the intention-to-treat (ITT) population who had no major protocol deviations. The ITT population is defined as all randomized subjects, analyzed according to their randomized treatment assignment.
Measure: Median (95% Confidence Interval); unit: Days to resolution of diarrhea
Arm/Group | Segment 2B: Ibezapolstat Arm--Double-blind, Randomized, Active-controlled Clinical Segment | Segment 2B: Vancomycin Arm--Double-blind, Randomized, Active-controlled Clinical Segment
Number analyzed (Participants) | 16 | 14
Days to resolution of diarrhea | 8 [4 to 10] | 9 [6 to 11]

13. Other Pre Specified Outcome: Segment 2A: Microbiome Effects
Description: The Shannon Diversity Index and Inverse Simpson Diversity Index are used to quantify biodiversity in a community like the gut microbiome, measuring how many different species are present in a community (richness) and how close in numbers different species in the community are to each other (evenness). The Shannon considers both factors while the Inverse Simpson focuses on evenness. The Shannon diversity index is calculated using natural logarithms, and units cancel out in the calculation, so it lacks units. It ranges from 0 to infinity. The Inverse Simpson represents the likelihood of selecting two different individuals from a population. It is a ratio and has no units. It ranges from 0 to 1. For both indexes, higher values indicate greater diversity.
Time Frame: Days 10 and 40
Population: 8 of the 10 participants in Segment 2A provided stool samples and were analyzed. Not all 8 subjects were able to provide samples for all time points, so the data are not continuous. Data is reported as mean increase in biodiversity from the baseline.
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | Segment 2A: Ibezapolstat (ACX-362E) Open-Label Single-Arm
Number analyzed (Participants) | 8
Index
  Change from Baseline on Inverse Simpson Index, during treatment (until Day 10) | 0.14 (0.06)
  Change from Baseline on Inverse Simpson Index, after treatment (until Day 40) | 0.22 (0.10)
  Change from Baseline on Shannon Diversity Index, during treatment (until Day 10) | 0.98 (0.48)
  Change from Baseline on Shannon Diversity Index, after treatment (until Day 40) | 1.7 (0.87)

14. Other Pre Specified Outcome: Segment 2B Per Protocol (PP) Population: Change From Baseline in EuroQoL 5 Dimension 5 Level (EQ-5D-5L) Quality of Life Scores
Description: Change from baseline in each of the 5 dimensions of the EQ-5D-5L score, each scored on a scale of 1-5, with 1 being normal and 5 indicating extreme difficulty or impairment. The 5 dimensions are mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Summary Index Scores (the 5 dimensions combined into a single value) are reported here. Values for the index score ranges from -0.59 to 1, where 1 is the best possible health state.
Time Frame: Days 12, 38, 66, and 94
Population: PP participants were those in the intent-to-treat (ITT) population who had no major protocol deviations. The ITT population is defined as all randomized subjects, analyzed according to their randomized treatment assignment.
Measure: Mean (Standard Deviation); unit: Summary Index Score
Arm/Group | Segment 2B: Ibezapolstat Arm--double-blind, Randomized, Active-controlled Clinical Segment | Segment 2B: Vancomycin Arm--double-blind, Randomized, Active-controlled Clinical Segment
Number analyzed (Participants) | 16 | 14
Summary Index Score
  Day 12 | 0.1667 (0.1226) | 0.1611 (0.1203)
  Day 38 | 0.1908 (0.1379) | 0.1897 (0.1506)
  Day 66: number analyzed (Participants) | 6 | 8
  Day 66 | 0.2677 (0.1649) | 0.1964 (0.1124)
  Day 94: number analyzed (Participants) | 6 | 8
  Day 94 | 0.2677 (0.1649) | 0.2004 (0.1158)

15. Other Pre Specified Outcome: Segment 2B Intent-to-Treat (ITT) Extension Population: Extended Clinical Cure (ECC) of Clostridioides Difficile Infection (CDI)
Description: Clinical cure (CC) at the test of cure (TOC) visit (ie, at least 48 hours after end of treatment [day 10]) and no recurrence within 56 days [day 66] or within 84 days [day 94]. Recurrence was defined as a new episode of diarrhea (3 or more UBMs in a 24-hour period) with a positive toxin result, using a Sponsor-approved C. difficile free toxin test and, in the opinion of the Investigator, requiring retreatment with an antibacterial agent for C. difficile.
Time Frame: 56 days after end of treatment (Day 66) and 84 days after end of treatment (Day 94)
Population: Participants from the ITT population were recruited for an extended follow-up period. In the ITT extension population, 1 ibezapolstat subject failed at the CC (Day 12) and 1 vancomycin subject failed at the SCC (Day 38); both failures carried forward to both ECC evaluations. There were no failures post SCC (Day 38). In the ITT extension population who achieved a SCC, 5/5 ibezapolstat-treated participants and 7/7 vancomycin-treated participants experienced no infection recurrence.
Measure: Count of Participants; unit: Participants
Arm/Group | Segment 2B: Ibezapolstat Arm--double-blind, Randomized, Active-controlled Clinical Segment | Segment 2B: Vancomycin Arm--double-blind, Randomized, Active-controlled Clinical Segment
Number analyzed (Participants) | 6 | 8
Participants
  Extended Clinical Cure 56 days after End of Treatment (Day 66): yes | 5 | 7
  Extended Clinical Cure 56 days after End of Treatment (Day 66): no | 1 | 1
  Extended Clinical Cure 84 days after End of Treatment (Day 94): yes | 5 | 7
  Extended Clinical Cure 84 days after End of Treatment (Day 94): no | 1 | 1

ADVERSE EVENTS:
Time Frame: 40 days--from the time the participant gave informed consent through study completion
Description: Participants were instructed to report AEs at each study visit. Study visits occurred on Days 1, 3, 5, 8, 10, 12, 20, 30, 38, and 40. No participants had AEs leading to study withdrawal or discontinuation.
Groups:
- Segment 2B: Ibezapolstat Arm--Double-blind, Randomized, Active-controlled Clinical Segment: Participants with diarrhea caused by C. difficile who were randomized to this arm received 450 mg ibezapolstat (3 x 150 mg capsules) every 12 hours for 10 days with placebo every 12 hours for 10 days (to maintain blind). Participants were followed for 28±2 days for recurrence. Blinding was maintained by over-encapsulation. 1 participant from the original population did not receive the study drug and was not included in calculations.
Arm/Group | Segment 2A: Ibezapolstat (ACX-362E) Open-Label Single-Arm | Segment 2B: Ibezapolstat Arm--Double-blind, Randomized, Active-controlled Clinical Segment | Segment 2B: Vancomycin Arm--Double-blind, Randomized, Active-controlled Clinical Segment
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/17 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/17 | 0/14
Other Adverse Events (participants affected / at risk) | 4/10 | 6/17 | 2/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Segment 2A: Ibezapolstat (ACX-362E) Open-Label Single-Arm (N=10) | Segment 2B: Ibezapolstat Arm--Double-blind, Randomized, Active-controlled Clinical Segment (N=17) | Segment 2B: Vancomycin Arm--Double-blind, Randomized, Active-controlled Clinical Segment (N=14)
Herpes zoster a (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Segment 2A: Ibezapolstat (ACX-362E) Open-Label Single-Arm (N=10) | Segment 2B: Ibezapolstat Arm--Double-blind, Randomized, Active-controlled Clinical Segment (N=17) | Segment 2B: Vancomycin Arm--Double-blind, Randomized, Active-controlled Clinical Segment (N=14)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Skin candida (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor is responsible for the conduct of the study, data analyses, and all results. All data are proprietary and belong to the sponsor, not to the investigator.

DOCUMENTS (2):
  • Study Protocol (2023-04-03): https://cdn.clinicaltrials.gov/large-docs/42/NCT04247542/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-25): https://cdn.clinicaltrials.gov/large-docs/42/NCT04247542/SAP_001.pdf